CLINICAL TRIAL: NCT04339933
Title: Detection of FGFR Gene Mutations in the Tumor Tissue and Urine of Patients With Urothelial Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ho Kyung Seo (Other Government)
Responsible Party: Sponsor-Investigator, Ho Kyung Seo, Senior Scientist, National Cancer Center, Korea
Organization: National Cancer Center, Korea (Other Government)
Other Study IDs: U-FGFR
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Study samples (8 ml blood and 20 ml urine) will be collected once within one month before treatment and once within three months after treatment, from the subjects who will agree to participate in the study.
  * Additional study samples will be collected once (8 ml blood and 20 ml urine) after surgery (or neoadjuvant chemotherapy).
  * Tissue samples will be collected during transurethral resection of bladder tumor (TUR-BT) before BCG therapy or after TUR-BT and cystectomy before and after neoadjuvant chemotherapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BC: Patients who were diagnosed with bladder cancer
  Interventions: Diagnostic Test: FGFR test

INTERVENTIONS:
Diagnostic Test: FGFR test — Detection of FGFR gene mutations in the tumor tissue and urine of patients

SUMMARY:
This study aims to compare the correlation between FGFR mutations found in bladder cancer tissues and urine to develop a companion diagnostic method for predicting the effect of FGFR inhibitors using urine samples of the patients with urothelial cancer.

DETAILED DESCRIPTION:
This study targets 92 patients with urothelial cancer, whose tissue (from scheduled surgery) and urine samples can be obtained, regardless of the treatment stage.

■ Examination Methods

* FGFR mutations in bladder cancer tissues will be analyzed using next-generation sequencing and current companion diagnostic methods.
* FGFR mutations in urine samples obtained from patients with bladder cancer will be analyzed using nanowires.
* Bladder cancer subtyping will be performed by RNA sequencing of tumor tissues or other methods.
* Analysis of paired tissues before and after chemotherapy will be performed on transurethral resection of bladder tumor (TUR-BT) and cystectomy tissues before and after neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Suspected patients of urothelial cancer who will visit the National Cancer Center Korea from the date of Institutional Review Board (IRB) approval to 2021 and with identified tumors in the bladder according to bladder endoscopy.
* Subjects who are scheduled for surgery (transurethral bladder tumor resection, radical bladder resection, and radical bladder ureterectomy) and have agreed to participate in the study

Exclusion Criteria:

* History of other active malignant tumors treated within 24 months
* Patients with either mental illness or who cannot participate in clinical trials at the judgment of other doctors
* If patients and guardians do not want to participate in this study
* History of having administered FGFR inhibitors in the past

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected patients of urothelial cancer who will visit the National Cancer Center Korea.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between FGFR mutations found in bladder cancer tissues and urine before and after treatment | Up to two weeks before and after surgery
  The ratio of patients with matching test results to total patients

SECONDARY OUTCOMES:
Changes in FGFR mutations in tissues before and after treatment | Up to two weeks before and after treatment
  Changes in FGFR mutations in tissues before and after treatment will be observed in the patients with muscle-invasive and non-muscle-invasive bladder cancer undergoing neoadjuvant chemotherapy and transurethral bladder tumor resection, respectively, due to recurrence.
Patient prognosis | six months and one year after treatment
  recurrence-free
Patient prognosis | six months and one year after treatment
  progression-free
Patient prognosis | six months and one year after treatment
  cancer-specific survivals
Patient prognosis | six months and one year after treatment
  overall survivals
PD-L1 expression | Up to two weeks before and after treatment
  PD-L1 expression level will be measured using immunohistochemistry, RNA sequencing, and other suitable methods to analyze the bladder cancer subtypes

CONTACTS AND LOCATIONS:
Overall Officials: Ho Kyung Seo, MD, PhD, Principal Investigator — National Cancer Center, Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cancer Genome Atlas Research Network. Comprehensive molecular characterization of urothelial bladder carcinoma. Nature. 2014 Mar 20;507(7492):315-22. doi: 10.1038/nature12965. Epub 2014 Jan 29. PMID 24476821
- [Background] Loriot Y, Necchi A, Park SH, Garcia-Donas J, Huddart R, Burgess E, Fleming M, Rezazadeh A, Mellado B, Varlamov S, Joshi M, Duran I, Tagawa ST, Zakharia Y, Zhong B, Stuyckens K, Santiago-Walker A, De Porre P, O'Hagan A, Avadhani A, Siefker-Radtke AO; BLC2001 Study Group. Erdafitinib in Locally Advanced or Metastatic Urothelial Carcinoma. N Engl J Med. 2019 Jul 25;381(4):338-348. doi: 10.1056/NEJMoa1817323. PMID 31340094
- [Background] Wu YM, Su F, Kalyana-Sundaram S, Khazanov N, Ateeq B, Cao X, Lonigro RJ, Vats P, Wang R, Lin SF, Cheng AJ, Kunju LP, Siddiqui J, Tomlins SA, Wyngaard P, Sadis S, Roychowdhury S, Hussain MH, Feng FY, Zalupski MM, Talpaz M, Pienta KJ, Rhodes DR, Robinson DR, Chinnaiyan AM. Identification of targetable FGFR gene fusions in diverse cancers. Cancer Discov. 2013 Jun;3(6):636-47. doi: 10.1158/2159-8290.CD-13-0050. Epub 2013 Apr 4. PMID 23558953